CLINICAL TRIAL: NCT03065829
Title: The Mediating Effects of Decentering on Self-Management Behaviors in Caregivers of Critically Chronically Ill Patients
Brief Title: Self-Management Behaviors of Caregivers of the Chronically Critically Ill
Acronym: ASSIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ronald Hickman, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11-15-11; P30NR015326 (NIH)
Record Dates: First submitted 2017-02-06; First posted 2017-02-28 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Critical Illness
Keywords: caregiver; chronically critically ill
MeSH Terms: conditions — Critical Illness | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Intervention Model Description: Our model posits that effective caregiver self-management depends on analytic and emotional processing. The investigators hypothesize the ASSIST intervention will improve analytic processing by improving self-monitoring. ASSIST will expose subjects to mindfulness meditation training and promote self-awareness, which will aid the regulation of their emotional processing and improve proximal outcomes. The investigators expect proximal self-management outcomes to influence the distal outcomes of caregiver health. Our model will also test the mediating effects of decentering, processing, the hypothalamic-pituitary axis (HPA), inflammatory stress response, and cognitive mediators. The influence of potential moderators will be assessed for their effect on the relationship between the self-management intervention and the proximal and distal outcomes.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASSIST (Experimental): The ASSIST intervention will deliver daily doses of MMT and vary dose intensity of all components each day based on the subject's biophysical data. Across a 30-day period, the ASSIST intervention will capture and analyze data to deliver on-demand MMT, guided practices to promote sleep hygiene and physical activity. Each day, subjects will receive at least one prompt to practice MMT (about 5 minutes at a time). However, based on the subject's biophysical sensor data, subjects could receive a maximum of 5 alerts or prompts per day from the device to enhance stress reduction, sleep hygiene, or physical activity.
  Interventions: Behavioral: ASSIST
- Attention-Control (Experimental): This intervention exposes subjects to the wearable technology without the self-management components to minimize novelty effects. Subjects assigned to this condition will wear the device for 30 days, which offers them an opportunity to experientially learn to self-monitor and employ self-regulatory skills by viewing the display biophysical data. Subjects in this condition will not receive any prompts from the device.
  Interventions: Behavioral: Attention-Control

INTERVENTIONS:
Behavioral: ASSIST — Wearable sensor technology delivering mindfulness meditation training (MMT) and health promotion (sleep hygiene and physical activity) .
  Arms: ASSIST
Behavioral: Attention-Control — Wearable sensor technology only viewing biophysical sensor data.
  Arms: Attention-Control

SUMMARY:
For family members of chronically critically ill (CCI) patients, an ICU admission marks a significant milestone in the patient's illness trajectory that highlights the onset of end of-life issues and an abrupt need for family members to assume the caregiver role for the first time. Assuming the caregiver role can have devastating and longstanding health consequences for family members, which can impair their ability to sustain caregiving behaviors for a CCI patient. The unrelenting psychological distress perceived by caregivers of CCI patients is linked to significant reductions in their self-management and health outcomes.

The purpose of this study is to evaluate a theoretically-derived Adaptive SenSor-Based Intervention for Caregiver Self-ManagemenT (ASSIST) intervention compared to an attention control condition for first time caregivers of CCI patients discharged to an extended care facility. One group will be exposed to the ASSIST intervention and will wear the sensor-based technology for 30 days and receive a daily dose of MMT. Biophysical sensor data (blood pressure, heart-rate variability, pedometry, and actigraphy) will be continuously acquired and analyzed using anomaly detection and machine learning techniques to vary the dose intensity (number of doses per day) of the two components of ASSIST adding a real-time, adaptive feature to promote caregiver self-management. The other group will wear the sensor-based technology for 30 days but will not receive the daily dose of MMT. The investigators will randomly assign participants to each group.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial to examine the ASSIST intervention compared to an attention control condition among 20 first time caregivers of CCI patients discharged to an extended care facility. The investigators will collect mixed methods data at baseline (T1) on Day 15 (T2) and Day 30 (T3) after subject enrollment to describe changes in proximal and distal outcomes. We have chosen our time points to capture neural and behavioral changes associated with the intervention.

The investigators aim to:

1. Determine whether there are differences in the distal outcomes [psychological burden (anxiety, depression, caregiver burden, HRQoL), cardiovascular health (BP and HRV) and economic costs] between subjects who were exposed to ASSIST compared to those exposed to the attention control condition.
2. Examine whether decentering, self-efficacy, decision-making, motivation, caregiver activation, and perceived stress mediate the relationship between exposure to a self-management condition (ASSIST vs. attention control) and the proximal (self-management) outcomes (stress reduction behaviors, sleep hygiene behaviors, and physical activity).
3. Determine if social support and demographics (gender and age) moderate the proximal outcomes [emotional distress, sleep quality, and physical activity] or distal outcomes [psychological burden (anxiety, depression, caregiver burden, HRQoL), cardiovascular health (BP and HRV) and economic costs].
4. Explore the differences in brain activation (structural and fMRI scans) and HPA function and stress response (hair cortisol, inflammation panel) between subjects exposed to ASSIST compared to those exposed to the attention control condition.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* recognized as the family member who will assume the caregiver role for a critically ill adult requiring at least 72 hours of mechanical ventilation and scheduled for a discharge to an extended care facility
* speak and comprehend English

Exclusion Criteria:

* currently practicing mindfulness-based interventions
* require psychotherapy or required psychotherapy within the last three months
* have a history of dementia or major neurological illness
* pregnant
* history of medical conditions or procedures that is contraindicated for fMRI scanning
* claustrophobia requiring anxiolytics or sedation
* expected to relocate from Northeast Ohio within two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Repeated Measures | Baseline to 30 days
  ANCOVA Model (F-Statistic)

SECONDARY OUTCOMES:
Change in Active Living Protocol (captured on wearable device) | From Baseline to up to 30 days
  Measure of Caregiver Sleep Activity
Change in Daily Diary of Physical Activity (captured on wearable device) | From Baseline to up to 30 days
  Measure of Caregiver Physical Activity
Change in Perceived Stress Scale | From Baseline to up to 30 days
  Measure of Caregiver Stress
Change in PROMIS-29 Scale | From Baseline to up to 30 days
  Measure of Caregiver Anxiety and Depression
Change in Zarits Burden Interview | From Baseline to up to 30 days
  Measure of Caregiver Burden
Change in Health Behaviors Questionnaire | From Baseline to up to 30 days
  Measure of Caregiver Health Related Quality of Life
Change in Heart Rate Variability (captured on wearable device) | From Baseline to up to 30 days
  Measure of Caregiver Heart Rate Variablity

CONTACTS AND LOCATIONS:
Overall Officials: Ronald L. Hickman, PhD, RN, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moore SM, Musil CM, Alder ML, Pignatiello G, Higgins P, Webel A, Wright KD. Building a Research Data Repository for Chronic Condition Self-Management Using Harmonized Data. Nurs Res. 2020 Jul/Aug;69(4):254-263. doi: 10.1097/NNR.0000000000000435. PMID 32205788